CLINICAL TRIAL: NCT03106259
Title: Observational Study to Evaluate the Safety of FURESTEM-RA Inj. in Moderate to Severe Rheumatoid Arthritis Patients Who Participated in Phase 1 Clinical Trial of FURESTEM-RA Inj
Brief Title: Long-term Observational Study to Evaluation the Safety of FURESTEM-RA Inj
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KSTBT_FURESTEM_RA_EXT
Record Dates: First submitted 2017-04-03; First posted 2017-04-10 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-08

CONDITIONS: Rheumatoid Arthritis
Keywords: FURESTEM-RA
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-Interventional Study: Subjects participating in this observational study originally participated in study FURESTEM-RA Inj.[NCT02221258]
  Interventions: Drug: FURESTEM-RA Inj.

INTERVENTIONS:
Drug: FURESTEM-RA Inj. — Non-interventional observational study
  Other Names: Not applicable-observational study

SUMMARY:
Observational Study to evaluate the safety of FURESTEM-RA lnj. in moderate to severe rheumatoid arthritis patients who participated in phase 1 clinical trial of FURESTEM-RA lnj.

DETAILED DESCRIPTION:
This is a observational study, single center, open label, study of safety of FURESTEM-RA Inj. in subjects with moderate to severe rheumatoid arthritis.

Subjects participating in this observational study originally participated in study FURESTEM-RA Inj.

[NCT02221258]

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in this observational study originally participated in study FURESTEM-RA Inj.[NCT02221258]
* Subject who understands and voluntarily sign an informed consent form

Exclusion Criteria:

* In case follow-up is not possible from end of clinical trial Phase 1 to end of this study period

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this observational study originally participated in study FURESTEM-RA Inj. [NCT02221258]
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2017-01-24 (Actual); Study Completion 2021-03-21 (Estimated)

PRIMARY OUTCOMES:
Safety of FURESTEM-RA Inj. | 5 years
  Evaluate the number of adverse events Safety of FURESTEM-RA Inj.

CONTACTS AND LOCATIONS:
Overall Officials: Ki-chul Shin, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul national University Boramae medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No